CLINICAL TRIAL: NCT01542645
Title: The Effect of Choice of Intraoperative Opioid on Postoperative Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Glenn Murphy, Director, Cardiac Anesthesia and clinical Research, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ENH10-256
Record Dates: First submitted 2012-02-26; First posted 2012-03-02 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Pain, Postoperative; Chronic Pain
Keywords: Fentanyl; Methadone; Thoracic Surgery
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain | interventions — Methadone; Analgesics, Opioid; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methadone (Experimental): Long-acting opioid
  Interventions: Drug: Methadone
- Fentanyl (Active Comparator): Shorter-acting opioid
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Methadone — Methadone (0.3 mg/kg) will be administered intraoperatively, with half of the dose given at induction of anesthesia (over 5 minutes) and the remainder administered as an infusion over the next 2 hours.
  Other Names: opioid
  Arms: Methadone
Drug: Fentanyl — Fentanyl (12 mcg/kg) will be administered intraoperatively, with half of the dose given at induction of anesthesia (over 5 minutes) and the remainder administered as an infusion over the next 2 hours.
  Other Names: opioid
  Arms: Fentanyl

SUMMARY:
The primary aim of this randomized, double-blind study is to examine the effect of a single intraoperative dose of methadone on postoperative pain and analgesic requirements in patients undergoing cardiac surgery with cardiopulmonary bypass. These patients will be compared to subjects receiving a standard dose of the "traditional" intraoperative opioid (fentanyl). Secondary outcome measures to be assessed will include standard recovery variables (such as length of postoperative intubation, ICU length of stay, incidence of nausea or vomiting, level of sedation). In addition, patients will be assessed for the development of chronic postoperative pain.

DETAILED DESCRIPTION:
Patients will be randomized to receive either methadone or fentanyl on the basis of a computer generated random number table. Patients in each group will receive standard intraoperative doses of either methadone or fentanyl that will allow for early tracheal extubation (within 4-8 hours of the conclusion of the surgical procedure). Study infusions will be prepared by the pharmacy, and all clinicians will be blinded to group assignment (methadone group-0.3 mg/kg-100 mL normal saline; fentanyl group-12 μg/kg-100 mL normal saline).

Pain will be assessed by blinded observers using a 11-point verbal analogue scale (0=no pain, 10=worst pain imaginable). Assessment for pain will be performed 15 minutes post-extubation and then 2, 4, 8, 12, 24, 48, and 72 hours after tracheal extubation. Pain will be determined at rest, with coughing, and during movement. At the same time pain data is collected, several other clinical assessments will be completed. The presence or absence of nausea and vomiting will be determined, and severity quantified using a 4-point ordinal scale (0=none, 3=severe). Level of sedation will be measured by observers using a 4-point sedation scale (0=fully awake, 1=mildly sedated (seldom drowsy and easy to awake), 2=moderately sedated (often drowsy and easy to awake), 3=severely sedated (somnolent, difficult to awake). Pruritis will also be measured using a 4-point scale (0=none, 3=severe). Any episodes of hypoventilation (respiratory rate < 8 breaths/min) or hypoxemia (oxygen saturation < 90%) during the study period will be recorded. Patient satisfaction with overall pain management will be determined using a 100-point verbal rating scale (1=highly dissatisfied (worst), 100=highly satisfied (best)). Respiratory rate, oxygen saturation (in ICU), and mean arterial blood pressure at the time of evaluation will be noted.

Postoperative pain will be managed according to standard institutional protocols. In the ICU, intravenous morphine will be administered for initial pain management (1 mg for mild-moderate pain, 2 mg for moderate-severe pain). Patients will be transitioned to oral pain medication when oral intake is tolerated (Norco tablets). The amount of pain medication administered during each study interval (listed above) will be recorded.

Other standard recovery variables will be recorded. These include time of initiation of ventilator weaning, time of tracheal extubation, arterial blood gas following extubation, time of ICU discharge, and time of hospital discharge. Time of first flatus and bowel movement will be recorded. Any complications during the hospitalization will be recorded. In a cohort of patients undergoing only coronary artery bypass graft surgery (n=75), serum troponins will be measured postoperatively to determine whether methadone has a potential cardioprotective effect.

Patients will be provided with a survey and self-addressed envelope following discharge from the hospital to determine the presence or absence of chronic persistent surgical pain. These data will be mailed by each patient 1, 3, 6, and 12 months postoperatively. The survey will assess the nature and severity of pain related to the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting for elective cardiac surgery with CPB will be eligible for enrollment.

Exclusion Criteria:

1. Preoperative renal failure requiring dialysis
2. Significant hepatic dysfunction (liver function tests > 2 times upper normal limit)
3. Preoperative ejection fraction < 30%
4. Pulmonary disease necessitating home oxygen therapy
5. Preoperative requirement for inotropic agents or intraaortic balloon pump to maintain hemodynamic stability
6. Allergy to methadone or fentanyl
7. Preoperative pain, use of preoperative opioids, or recent history of opioid abuse

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2010-09; Primary Completion 2013-11 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn S. Murphy, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Methadone | Fentanyl
Started | 82 | 82
Completed | 77 | 79
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methadone | Fentanyl | Total
Number analyzed (Participants) | 77 | 79 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (10.5) | 65.5 (11.1) | 65.1 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 16 | 41
  Male | 52 | 63 | 115

OUTCOME MEASURES:

1. Primary Outcome: Total Opioid Consumption in the Postoperative Period
Description: Total intravenous morphine used first three days (72 hours after ICU admission)
Time Frame: First 3 days after surgery
Measure: Median (Full Range); unit: milligrams
Arm/Group | Methadone | Fentanyl
Number analyzed (Participants) | 77 | 79
milligrams | 8 [0 to 44] | 14 [2 to 146]

2. Secondary Outcome: Postoperative Pain Scores
Description: Pain was assessed on a 11-point verbal analogue scale with 0=no pain, 10=worst pain imaginable
Time Frame: 2 hours after cardiac surgery
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Methadone | Fentanyl
Number analyzed (Participants) | 77 | 79
units on a scale | 3 [0 to 8] | 4.5 [0 to 10]

3. Secondary Outcome: Chronic Postoperative Pain Scores-Weekly Frequency of Pain
Description: 0=< once per week; 1=once per week; 2=twice per week; 3=daily; 4=constant
Time Frame: 1 months after surgery
Population: A home postal survey was sent to participants in the clinical trial 1 month after surgery. 46 patients in the methadone group and 58 patients in the fentanyl group returned the surveys
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Methadone | Fentanyl
Number analyzed (Participants) | 46 | 58
score on a scale | 0 [0 to 2] | 2 [0 to 3]

4. Secondary Outcome: Marker of Myocardial Injury (Troponin I)
Description: In a cohort of patients undergoing only coronary artery bypass graft surgery (n=75), serum troponins will be measured postoperatively to determine whether methadone has a potential cardioprotective effect.
Time Frame: 12 hours after surgery
Measure: Median (Full Range); unit: nanograms per millimeter
Arm/Group | Methadone | Fentanyl
Number analyzed (Participants) | 34 | 41
nanograms per millimeter | 5.4 [0.001 to 11.7] | 4.6 [0.7 to 30.0]

5. Secondary Outcome: 3 Months-Chronic Pain-weekly Frequency of Pain
Description: 0=< once per week; 1=once per week; 2=twice per week; 3=daily; 4=constant
Time Frame: 3 months
Population: A home postal survey was sent to participants in the clinical trial 3 months after surgery. 46 patients in the methadone group and 54 patients in the fentanyl group returned the surveys
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Methadone | Fentanyl
Number analyzed (Participants) | 46 | 54
score on a scale | 0 [0 to 2] | 0.5 [0 to 3]

6. Secondary Outcome: 6 Months-Chronic Pain-weekly Frequency of Pain
Description: 0=< once per week; 1=once per week; 2=twice per week; 3=daily; 4=constant
Time Frame: 6 months
Population: A home postal survey was sent to participants in the clinical trial 6 months after surgery. 42 patients in the methadone group and 39 patients in the fentanyl group returned the surveys
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Methadone | Fentanyl
Number analyzed (Participants) | 42 | 39
score on a scale | 0 [0 to 1] | 0 [0 to 1]

7. Secondary Outcome: 12 Months-Chronic Pain-weekly Frequency of Pain
Description: 0=< once per week; 1=once per week; 2=twice per week; 3=daily; 4=constant
Time Frame: 12 months
Population: A home postal survey was sent to participants in the clinical trial 12 month after surgery. 31 patients in the methadone group and 34 patients in the fentanyl group returned the surveys
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Methadone | Fentanyl
Number analyzed (Participants) | 31 | 34
score on a scale | 0 [0 to 0] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Methadone | Fentanyl
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/79
Other Adverse Events (participants affected / at risk) | 0/77 | 0/79

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No